CLINICAL TRIAL: NCT06127121
Title: A Digital Art Activity to Enhance Self-Disclosure and the Detection of Psycho-social Distress in Adult Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0328; NCI-2023-09557 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Digital Art Activity: Visit 1, Participants will be asked to complete a symptom questionnaire and then you will interact with the digital art tool. Participants will first complete a short breathing exercise, and then Participants will interact with the digital art tool. The digital tool combines a digital canvas with a collage activity. Participants will be asked to choose a background and then answer questions about your general well-being and your physical and emotional symptoms as they relate to cancer and cancer treatment.
  Visit 2, Participants will be asked to fill out the symptom questionnaire, complete another activity such as listening to meditative music for 10 minutes, and then fill out the symptom questionnaire again.
  Visit 3, Participants will fill out the symptom questionnaire and engage in the digital art activity again. Participants will then be asked to fill out 3 other questionnaires about your feelings of distress.
  Interventions: Behavioral: Digital Art Activity

INTERVENTIONS:
Behavioral: Digital Art Activity — * complete a symptom questionnaire
  * complete another activity such as listening to meditative music for 10 minutes
  * fill out the symptom questionnaire and engage in the digital art activity again

SUMMARY:
To look at how a digital art activity may help cancer patients improve their ability to express their distress, symptoms, and lived experience.

DETAILED DESCRIPTION:
Primary objective:

* To evaluate how engaging in a digital art activity might potentially cause changes in symptom reporting, based on pre/post self-reporting on the Edmonton Symptom Assessment System (ESAS) at time T3.

Secondary objectives:

* To evaluate the changes in symptom reporting, based on pre/post self-reporting on ESAS at different times of the study (T1, T2).
* To evaluate how a specific creative art making activity (T3), compared to an active control condition (T2; music listening) may or may not impact reporting ESAS.
* To monitor potential changes in distress disclosure, based on the self-report scoring on the Distress Disclosure Index score at T0, T2 and T3.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal or greater than 18 years
2. Patients who are admitted in the hospital and have received a cancer diagnosis.
3. Suffering from solid cancer or hematological malignancy and receiving active treatment for their cancer.
4. Voluntary written consent.
5. Fluent in English or Spanish.

Exclusion Criteria:

1. Not being able to use a digital tablet
2. Being speech impaired or vision impaired
3. Patients who are cognitively impaired and unable to read or consent for the study
4. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer Center
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
The Edmonton Symptom Assessment System, (ESAS) questionnaires | through study completion; an average 1 year.
  Score Scale (0-10) 0 No symptom-10 Worst possible

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Roldan, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org